CLINICAL TRIAL: NCT06583733
Title: On Any Page, Select Quit to Stop Entering Data. Data Entered on Previous Pages Will be Retained: To Complete Data Entry Later, Open the Record From the Home Page
Brief Title: Keep On Keep Up Bladder Health: Co-creating and Testing a Self-management Technological Solution for Ageing Well
Acronym: KOKU Bladder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: Hospital Universitari Santa Maria de Lleida (GSS) (Unknown); Institut de Recerca i Innovació en Ciències de la Vida i de la Salut a la Catalunya Central (IRIS) (Unknown); University of Manchester (Other); Research Council of Lithuania (Other); Lithuanian Sports University (Other); Agencia Gestió Ajuts Universitaris i Recerca (Unknown); Consorci Hospitalari de Vic (CHV) (Unknown)
Responsible Party: Principal Investigator, Javier Jerez Roig, Professor, Head of research group on Methodology, Methods, Models and Outcomes of Health and Social Science (M3O), University of Vic - Central University of Catalonia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOKU Bladder
Record Dates: First submitted 2024-09-01; First posted 2024-09-04 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Urinary Incontinence in Old Age
Keywords: pelvic health; urinary incontinence; aged; eHealth; behavior change; physical activity; sedentary behavior; bladder health; technology
MeSH Terms: conditions — Urinary Incontinence; Motor Activity; Sedentary Behavior | interventions — Health Planning Guidelines

STUDY DESIGN:
Intervention Model Description: 120 individuals will be simple randomised to a control (recommendations for self- managing urinary symptoms) or intervention (KOKU Bladder) group. It is anticipated that the multicomponent intervention will last 12 weeks and consist of health education, pelvic floor muscle exercises and BC techniques but this may vary according to the co-creation process. Measures will be assessed at baseline and end of intervention.
Masking Description: Usually, in physiotherapist studies it is very difficult to do blinding, because the patients can do some physical activity or exercise. In this trial, participants blinding will not be possible because the patients know what treatment they do, they should do the different exercises with app or with a HB information. Also, it is necessary to do face-to-face assessment for the physiotherapist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): The control group which will receive recommendations for self- managing urinary symptoms.
  There will be at least 60 participants (men and women mixed) distributed in 3 countries. It is anticipated that the multicomponent intervention will last 12 weeks.
  After the intervention we will collect the results with a mixed (qualitative and quantitative) approach.
  Interventions: Behavioral: recommendations
- intervention group (Experimental): The intervention group, which will receive the treatment with KOKU Bladder. There will be at least 60 participants (men and women mixed) distributed in 3 countries. It is anticipated that the multicomponent intervention will last 12 weeks.
  After the intervention we will collect the results with a mixed (qualitative and quantitative) approach.
  Interventions: Behavioral: KOKU Bladder

INTERVENTIONS:
Behavioral: KOKU Bladder — In this intervention the participants will receive treatment with the KOKU app ( based digital health program with behavior change techniques to improve bladder health ) for 12 weeks.
  After the intervention we will collect the results with a mixed (qualitative and quantitative) approach. Qualitative information will be recorded and analysed through thematic analysis, and quantitative data will be collected with tests and questionnaires.
  Arms: intervention group
Behavioral: recommendations — In this intervention the participants will receive recommendations for self- managing urinary symptoms, which they must follow for 12 weeks.
  After the intervention we will collect the results with a mixed (qualitative and quantitative) approach. Qualitative information will be recorded and analysed through thematic analysis, and quantitative data will be collected with tests and questionnaires.
  Arms: control group

SUMMARY:
KOKU Bladder aims to develop and test an evidence based digital health program with behavior change techniques to improve bladder health of adults aged 50 and over. A novel module embedded in the approved app "Keep-on-Keep-up" (KOKU) will be co-created with end-users, researchers, health professionals, and stakeholders through a participatory and appreciative action and reflection methodology. After a comprehensive literature review and consultation with 4-6 experts, 6 focus groups will be undertaken in Kaunas(Lithuanian), Catalonia (Spain) and Manchester (UK) to co-create the contents of the module. Data will be analyzed using thematic analysis. Gamification and the Honeycomb model for user experience will be followed to achieve an appropriate technological solution that will be tested through a randomized controlled trial with at least 120 individuals. A mixed methods approach (quantitative/qualitative analysis) will be used to assess the feasibility and acceptability of the program. Open data and science, gender and ethical aspects, as well as a risk management plan are considered. A plan for communication, dissemination, exploitation of results will be considered. KOKU Bladder will be highly scalable and will have wide reach and impact. This proposal is in line with EU policy initiatives on Active and Healthy Ageing (bladder health and continence will be promoted), targeting aspects such as eHealth, Innovation and Digital Care Transformation, by supporting users to demand more responsive and integrated care programs for chronic conditions and enhancing self-management strategies, independence and health intelligence.

DETAILED DESCRIPTION:
Phase I (month-M1-3): Prepare and submit protocol to Ethics Committee, conduct an updated review of the on eHealth solutions to manage UI using BCTs (e.g. training, education) that have been designed or tested in older adults, and establish contact with the Lithuanian, Spanish and UK participating institutions. Phase1 is dedicated to the management of the project throughout its duration.

Phase II (M2-5): Consultation with 4-6 experts on Badder Health (BH) and/or behavioral interventions. Develop a first iteration of the eHealth method and module.

Conduct an initial online focus group with 10-12 co-creators of UK to explore their perceived acceptability and feasibility and preferences for the eHealth program (concept development through co-creation).

Develop a first iteration of the eHealth method and module (concept development) - by Reason Digital (tech company in Manchester)

Phase III (M6-14): Organize, conduct and analyze 5 more focus group (2 in Lithuania, 1 UK and 2 Spain) with 10-12 co-creators each (community-dwelling people aged 50+ of both genders with different physical conditions and UI, health professionals and stakeholders with different backgrounds) to explore their perceived acceptability and feasibility and preferences for the eHealth program (concept development through co-creation). Secondment in University of Manchester.

Phase IV (M14-M20): Further develop the eHealth module (concept development) - by Reason Digital (tech company in Manchester)

Phase V (M21-36): Multicenter two-armed feasibility RCT study with at least 120 participants (WP3). Participants will be randomized to a control (recommendations for self- managing urinary symptoms) or intervention (KOKU Bladder) group.

Phase VI: Early and open communication and dissemination (WP4). Analysis of results.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 (range used in the literature covering the late-life process, including prostate issues and the perimenopause period)
* Self-reported UI (at least 1 leakage/month)
* Ability to read and understand the national languages
* Have a mobile phone/tablet
* Sign informed consent.

Exclusion Criteria:

* Red-flag symptoms (e.g., bleeding)
* Unstable health conditions.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
To co-create, develop and test an evidence based digital health program with behavior change techniques to decrease UI of community-dwelling adults aged 50 and over | 3 years
  The primary aim of KOKU Bladder is to co-create and test an eHealth program to address bladder health (specifically urinary incontinence) in community-dwelling adults aged 50 and over

SECONDARY OUTCOMES:
To evaluate the life-impact related to UI (Incontinence Impact Questionnaire-7) of community-dwelling adults aged 50 and over. | 3 years
  We will use the Incontinence Impact Questionnaire-7 (IIQ-7) to assess it
To evaluate the lower urinary tract symptoms (International Prostate Symptom Score) of community-dwelling adults aged 50 and over. | 3 years
  We will use different questionnaires.
To evaluate the Patient Global Impression of Improvement; SB (visual analogue scale, a 7-day recall period) of community-dwelling adults aged 50 and over | 3 years
  We will use a visual analogue scale to assess it
To evaluate the satisfaction with treatment of community-dwelling adults aged 50 and over. | 3 years
  We will use different questionnaires.
To modify the severity of UI (International Consultation on Incontinence Questionnaire-UI short form) of community-dwelling adults aged 50 and over | 3 years
  We will use the International Incontinence Questionnaire-Short Form (ICIQ-SF) to assess it

CONTACTS AND LOCATIONS:
Overall Officials: Jerez-Roig, PhD, Principal Investigator — University of Vic-Central University of Catalonia; Lithuanian Sports University
Locations (4):
- Lithuanian Sports University, Kaunas, Lithuania
- Spain (2):
  - Hospital Santa Maria, Lleida
  - Hospital Consortium of Vic, Vic
- University of Manchester, Manchester, United Kingdom

REFERENCES:
- [Derived] Jerez-Roig J, Aguila-Gimeno O, Brazaitis M, Solianik R, Karkauskiene E, Jarutiene L, Fuente-Vidal A, Borralleras-Fumana E, Gasteiger N, Stanmore E. Co-creating and testing a self-management digital solution for bladder health and urinary continence among people aged 50 and over: protocol for the international KOKU Bladder project. BMJ Open. 2025 Sep 11;15(9):e100487. doi: 10.1136/bmjopen-2025-100487. PMID 40940057